CLINICAL TRIAL: NCT03057912
Title: A Safety and Efficacy Study of Transcription Activator-like Effector Nucleases and Clustered Regularly Interspaced Short Palindromic Repeat/Cas9 in the Treatment of HPV-related Cervical Intraepithelial NeoplasiaⅠ
Brief Title: A Safety and Efficacy Study of TALEN and CRISPR/Cas9 in the Treatment of HPV-related Cervical Intraepithelial NeoplasiaⅠ
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Jingchu University of Technology (Other)
Responsible Party: Principal Investigator, Hu Zheng, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017CRISPR/Cas9&TALEN
Record Dates: First submitted 2017-02-12; First posted 2017-02-20 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Human Papillomavirus-Related Malignant Neoplasm
Keywords: Cervical intraepithelial neoplasiaⅠ; TALEN; CRISPR/Cas9
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Transcription Activator-Like Effector Nucleases; CRISPR-Associated Protein 9

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TALEN (Experimental): TALEN (TALEN-HPV16 E6/E7 or TALEN-HPV18 E6/E7) plasmid in gel, administered twice one week for 4 weeks.
  Interventions: Biological: TALEN
- CRISPR/Cas9 (Experimental): CRISPR/Cas9 (CRISPR/Cas9-HPV16 E6/E7T1 or CRISPR/Cas9-HPV18 E6/E7T2 ）plasmid in gel, administered twice one week for 4 weeks.
  Interventions: Biological: CRISPR/Cas9
- Control group (No Intervention): Observation

INTERVENTIONS:
Biological: TALEN — TALEN gel consists of TALEN plasmid, C32-447, Poloxmer 407 and distilled water as solvent.
  Other Names: TALEN-HPV16 E6/E7;TALEN-HPV18 E6/E7
  Arms: TALEN
Biological: CRISPR/Cas9 — CRISPR/Cas9 gel consists of CRISPR/Cas9 plasmid, C32-447, Poloxmer 407 and distilled water as solvent.
  Other Names: CRISPR/Cas9-HPV16 E6/E7T1;CRISPR/Cas9-HPV18 E6/ E7T2
  Arms: CRISPR/Cas9

SUMMARY:
This is an open-label and triple cohort study of the safety and efficacy of TALEN and CRISPR/Cas9 to possibly treat HPV Persistency and human cervical intraepithelial neoplasiaⅠwithout invasion.

DETAILED DESCRIPTION:
HPV persistent infection is the major causal factor of cervical intraepithelial neoplasia (CIN) and cervical cancer. The important roles of E6 and E7 playing in HPV-driven carcinogenesis make them attractive targets for therapeutic interventions. Previous evidences showed that using designated TALEN and CRISPR/Cas9 as genome editing tool could produce disruption of HPV16 and HPV18 E6/E7 DNA, significantly decreasing the expression of E6/E7, inducing cell apoptosis and inhibiting cell lines growth.

This study will evaluate the safety and efficacy of TALEN-HPV E6/E7 and CRISPR/Cas9-HPV E6/E7 in treating HPV Persistency and HPV-related Cervical Intraepithelial NeoplasiaⅠ

ELIGIBILITY:
Inclusion Criteria:

* Documented HPV16 or HPV18 infection.
* Married and fertile, no fertility requirements.
* Without administration of hormone in the last six months.
* Subjects must be meet the ethical requirements and have signed informed consent.

Exclusion Criteria:

* Pregnancy and breast feeding
* Any bacterial vaginitis
* Any Fungal vaginitis
* Any sexually transmitted diseases
* Active drug or alcohol abuse
* Any HPV medications within the past 12 weeks
* Allergy to active or non active ingredients in the study of drugs
* Cardiac insufficiency
* Liver and renal insufficiency
* Hypertension and severe complications
* Serious illness in past 30 days
* Currently participating in another clinical trial or any prior gene therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-11-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 6 months
  The primary objective of this Study is to evaluate the safety of therapeutic doses and the dosing regimen of TALEN and CRISPR/Cas9 plasmid.

SECONDARY OUTCOMES:
Change of HPV16 or 18 DNA titers | Baseline, 3 and 6 months
  Blood samples will be taken at the baseline, months 3 and 6 on each subject.
Change of cervical cytological results. | Baseline, 3 and 6 months
  ThinPrep Pap Test will be conducted at the baseline, months 3 and 6 on each subject.
Change of cervical histological results. | Baseline and 6 months.
  Colposcopy Biopsy will be conducted at the baseline and month 6 on each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Hu, M.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hu Z, Yu L, Zhu D, Ding W, Wang X, Zhang C, Wang L, Jiang X, Shen H, He D, Li K, Xi L, Ma D, Wang H. Disruption of HPV16-E7 by CRISPR/Cas system induces apoptosis and growth inhibition in HPV16 positive human cervical cancer cells. Biomed Res Int. 2014;2014:612823. doi: 10.1155/2014/612823. Epub 2014 Jul 20. PMID 25136604
- [Background] Hu Z, Ding W, Zhu D, Yu L, Jiang X, Wang X, Zhang C, Wang L, Ji T, Liu D, He D, Xia X, Zhu T, Wei J, Wu P, Wang C, Xi L, Gao Q, Chen G, Liu R, Li K, Li S, Wang S, Zhou J, Ma D, Wang H. TALEN-mediated targeting of HPV oncogenes ameliorates HPV-related cervical malignancy. J Clin Invest. 2015 Jan;125(1):425-36. doi: 10.1172/JCI78206. Epub 2014 Dec 15. PMID 25500889